CLINICAL TRIAL: NCT02099552
Title: Natural History and Outcomes in X-Linked Hypohidrotic Ectodermal Dysplasia
Acronym: ECP-015
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-015
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: X-Linked Hypohidrotic Ectodermal Dysplasia
Keywords: X-Linked hypohidrotic ectodermal dysplasia; XLHED; Hypohidrotic ectodermal dysplasia; HED; Christ-Siemens-Touraine syndrome
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- XLHED: Those with the condition of XLHED

SUMMARY:
The proposed natural history study will enroll male and female patients, ages 36 months and younger, who have a diagnosis of XLHED based on genetic testing and who have not received an investigational study drug. The study protocol will include collection of all relevant medical history and documentation of clinical outcomes using age-appropriate, minimally invasive technologies. Data will be collected both retrospectively, back to pregnancy assessments that may be available, and prospectively through age 5 yrs.

DETAILED DESCRIPTION:
Important to the development and regulatory approval of therapies for XLHED will be the collection of data on the clinical history and prospective health of those affected by XLHED. The proposed natural history study will enroll male and female patients, ages 36 months and younger, who have a diagnosis of XLHED based on genetic testing and who have not received an investigational study drug. The study protocol will include collection of all relevant medical history and documentation of clinical outcomes using age-appropriate, minimally invasive technologies. Data will be collected both retrospectively, back to pregnancy assessments that may be available, and prospectively through age 5 yrs. Genotype-phenotype correlations in XLHED, based on well-documented health records and prospective assessments on genetically-confirmed individuals, may now provide new and clinically-predictive information for the benefit of patients, families, health care providers and clinical investigators designing trials for therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled in this study:

1. Confirmed genetic diagnosis of XLHED
2. Written informed consent of both parents (if reasonably available)

Exclusion Criteria:

Subjects who meet any of the following criteria cannot be enrolled in this study:

1. Medically-significant complications or congenital anomalies outside of those considered to be associated with the diagnosis or status of XLHED
2. Having received an investigational study drug prior to enrollment. For subjects less than 6 months of age, the mother cannot have taken an investigational drug during her pregnancy.
3. Known hypersensitivity to pilocarpine or pilocarpine-like muscarinic agonists
4. Presence of pacemakers

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Those with the condition of XLHED up to age 36 months
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To assess clinical course of untreated XLHED individuals | Up to 5 years of life
  To characterize the clinical course of untreated XLHED male and female subjects in early childhood, capturing data from physician and hospital records, medical history including growth and development, and family interviews.
To assess the phenotype of untreated XLHED individuals | Up to 5 years of life
  To characterize the phenotype of untreated XLHED male subjects and female in early childhood with endpoint assessments including sweat (males only), dentition, craniofacial development, pulmonary and ocular health.

SECONDARY OUTCOMES:
To assess changes in endpoint assessments over time (growth and development) | Baseline and yearly up through 5 years of age
To assess changes in endpoint assessments over time (Mortality/Hospitalizations/Infections/Fevers/Heat Intolerance) | Baseline and yearly up through 5 years of age
To assess changes in endpoint assessments over time (sweat rate) | Baseline and yearly through 5 years of age
To assess changes in endpoint assessments over time (Dentition) | Baseline and yearly through 5 years of age
To assess changes in endpoint assessments over time (dry eye) | Baseline and yearly through 5 years of age
To assess changes in endpoint assessments over time (skin, hair and nail health) | Baseline through 5 years of age
To assess changes in endpoint assessments over time (respiratory health) | Baseline and yearly through 5 years of age
To assess changes in endpoint assessments over time (craniofacial development) | Baseline and yearly through 5 years of age
To assess genotype-phenotype correlation in XLHED affected individuals | Baseline through 5 years of age
  To correlate clinical course and endpoint outcomes with EDA genotype in untreated XLHED-affected male and female subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ramsey Johnson, MSM, Study Director — Edimer Pharmaceuticals
Locations (7):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University School of Medicine, St Louis, Missouri
- Hôpital Necker-Enfants Malades, Paris, France
- University Hospital Erlangen, Erlangen, Bavaria, Germany
- Azienda Ospedaliera-Polo Universitario "Luigi Sacco", Milan, Italy
- University Hospital of Wales, Cardiff, United Kingdom